CLINICAL TRIAL: NCT02892578
Title: Systematic Screening With Electrocardiogram for Unknown Atrial Fibrillation in 65 Years Old and Above People in Nursing Home
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Study halted prematurely because the potential for recruitment into the associated center was reached.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9581
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- electrocardiogram (Experimental): Patient will take an electrocardiogram in order to detect atrial fibrillation
  Interventions: Other: electrocardiogram

INTERVENTIONS:
Other: electrocardiogram

SUMMARY:
Atrial fibrillation is the most common arrhythmia. Some studies shown that systematic screening with electrocardiogram could improve atrial fibrillation detection. No studies are available in nursing home. The goal of this study is to screen atrial fibrillation in patients who live in nursing home.

DETAILED DESCRIPTION:
A prospective observational cross sectional multicenter study.

The goal of this study is to detect atrial fibrillation in nursing home people aged 65 years old and above, with systematic electrocardiogram. Participants agreement will be collected. Participants characteristics data will be collected in all nursing home. For all participants, one visit were realised with electrocardiogram, and symptoms survey. Data were anonymised on each center before analysed.

ELIGIBILITY:
Inclusion criteria :

* Being in nursing home since 1 month and above
* Aged > 65 years old
* Subjects agree to participate at this project

Exclusion criteria :

* Antecedent of atrial fibrillation

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 287 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
presence of atrial fibrillation on electrocardiogram | up to 1 hour
  detection of atrial fibrillation during the electrocardiogram

SECONDARY OUTCOMES:
presence of irregular pulse | up to 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Heart and vascular diseases service, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided